CLINICAL TRIAL: NCT03897933
Title: Erector Spinae Plane Block for Postoperative Pain in Percutaneous Nephrolithotomy Patients: a Retrospective Study
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sibel Seçkin Pehlivan, Teaching Assistant, TC Erciyes University
Other Study IDs: 2019/881
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2020-01

CONDITIONS: Percutaneous Nephrolithotomy
Keywords: Erector spinae block; percutaneous; nephrolithotomy; stone; ultrasound
MeSH Terms: conditions — Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Erector spinae plane block group (ESP): Single- shot ultrasound guided ESP block with 30 ml 0.25% bupivacain at the T10 vertebral level was performed preoperatively to patients in the ESP group (Group I).
  Interventions: Procedure: Erector Spinae Plane block ( Group I)
- non- blocked Group: consists of the patient group without any procedure
  Interventions: Procedure: non- blocked Group (GROUP II)

INTERVENTIONS:
Procedure: Erector Spinae Plane block ( Group I) — ESP Block was performed preoperative to all patients in ESP block group. Patients in all groups were provided with intravenous patient- controlled analgesia device containing morphine for postoperative analgesia.
  Groups: Erector spinae plane block group (ESP)
Procedure: non- blocked Group (GROUP II) — This group was received no intervetion. Patients in all groups were provided with intravenous patient- controlled analgesia device containing morphine for postoperative analgesia.
  Groups: non- blocked Group

SUMMARY:
To evaluate the ability of Erector spina Plane block decrease postoperative pain and analgesia requirements in patients undergoing Percutaneous Nephrolithotomy.

DETAILED DESCRIPTION:
Erector spina Plane block was performed with guided ultrasound at T10 Transverse process level would lead to adequate postoperative analgesia ,in Percutaneous Nephrolithotomy surgeries.

ELIGIBILITY:
Inclusion Criteria:

* ASA I- ASA II Patients

Exclusion Criteria:

* history of allergy to the study medication
* refusal to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A number of 60 patients undergoing PCNL between January 2019 and December 2019 were included in our study. Patients included in the study were those who were operated from the stone diseases.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
opioid consumption | 24 hours after surgery
  In the recovery room, all patients were given a patient- controlled analgesia device containing morphine 0.5 mg/ml, set to deliver a 1mg bolus dose of morphine with an 10 min lockout time and 10 mg 4 h limit.Total morphine consumption during the 24 hours postoperative period will recorded at 5 times intervals ( 2, 4, 6, 12, 24 hours).
Verbal analog Pain Scores on rest and movement | 24 hours after surgery
  A Research assistant, blinded to the group allocation, interviewed patients and collected data at 5 times intervals ( 2, 4, 6, 12, 24, hours) in the 24 hours postoperatively. Patients were asked to rate their pain using verbal analog scale, where 0= no pain and 10= worst pain possible.

SECONDARY OUTCOMES:
Demographic data | 24 hours after surgery
  Age, BMI, ASA, Duration of surgery was recorded.
incidences of adverse effects (like nausea and vomiting) | 24 hours after surgery
  incidences of nausea and vomiting during the 24 hours postoperative period was recorded recorded at 5 times intervals ( 2, 4, 6, 12, 24 hours).

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Pehlivan, Study Director — TC Erciyes University
Locations (1):
- Sibel Seçkin Pehlivan, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 24 months of study completion
Access Criteria: Data accept requests will be reviewed by an external independent Review Panel.Requesters will be required to sign a Data Access Agreement

REFERENCES:
- [Result] Liu X, Huang G, Zhong R, Hu S, Deng R. Comparison of Percutaneous Nephrolithotomy Under Regional versus General Anesthesia: A Meta-Analysis of Randomized Controlled Trials. Urol Int. 2018;101(2):132-142. doi: 10.1159/000491021. Epub 2018 Jul 20. PMID 30032149
- [Result] Elkassabany N, Ahmed M, Malkowicz SB, Heitjan DF, Isserman JA, Ochroch EA. Comparison between the analgesic efficacy of transversus abdominis plane (TAP) block and placebo in open retropubic radical prostatectomy: a prospective, randomized, double-blinded study. J Clin Anesth. 2013 Sep;25(6):459-65. doi: 10.1016/j.jclinane.2013.04.009. Epub 2013 Aug 17. PMID 23965191
- [Result] Gurkan Y, Aksu C, Kus A, Yorukoglu UH, Kilic CT. Ultrasound guided erector spinae plane block reduces postoperative opioid consumption following breast surgery: A randomized controlled study. J Clin Anesth. 2018 Nov;50:65-68. doi: 10.1016/j.jclinane.2018.06.033. Epub 2018 Jul 2. PMID 29980005